CLINICAL TRIAL: NCT04736108
Title: A Single-center, Phase II Neoadjuvant Study of Abiraterone Acetate in the Treatment of Intraductal Carcinoma of the Prostate
Brief Title: Neoadjuvant Therapy of Abiraterone Plus ADT for Intraductal Carcinoma of the Prostate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Professor of Department of Urology, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201224; Dragon-001 (Other: Chia Tai Tianqing Pharmaceutical Group Co., LTD)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: abiraterone acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisolone; Goserelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADT with Abiraterone and prednisone (Experimental): All subjects in this arm will receive luteinizing hormone releasing hormone analogue (LHRHa) plus abiraterone acetate and prednisone, as per standard of care. Goserelin 10.8 mg will be used once per 12 weeks. Abiraterone acetate will be administered orally as 1000 mg once daily along with 5 mg of oral prednisone once per day. Subjects will continue to take abiraterone acetate and prednisone for 24 weeks before radical prostatectomy
  Interventions: Drug: Abiraterone acetate; Drug: Prednisolone; Drug: Goserelin

INTERVENTIONS:
Drug: Abiraterone acetate — 1000 mg orally daily for 24 weeks before radical prostatectomy
Drug: Prednisolone — 5 mg oral low dose prednisone, once daily
Drug: Goserelin — 10.8 mg goserelin hypodermic once per 12 weeks

SUMMARY:
Neoadjuvant treatment before radical prostatectomy has been proven to provide benefits on peri-operation results, especially on reduction of tumor volume and minimization of biochemical recurrence. This study will evaluate the efficacy and safety of abiraterone acetate Plus androgen deprivation therapy（ADT）in high-risk localized prostate cancer with intraductal carcinoma of the prostate（IDC-P）.

DETAILED DESCRIPTION:
IDC-P is an adverse pathological entity of prostate cancer, characterized by the growth of malignant cells in pre-existing prostatic ducts and acini, and is present in high-grade disease and associated with poor prognosis. Previous studies have shown that IDC-P was significantly associated with an adverse clinical course in patients who received radical prostatectomy or radiotherapy, and the presence of IDC-P on the biopsy specimen was associated with a poor prognosis in terms of overall survival (OS) and a poor docetaxel response in patients with distant metastasis at the initial diagnosis. Our previous researches as well as other published data indicated that abiraterone had a better therapeutic efficacy than docetaxel as the first-line therapy in metastatic castration resistance prostate cancer（mCRPC）with IDC-P. Therefore we intended to perform this single-arm phase II clinical trial to evaluate the initial efficacy and safety of abiraterone acetate Plus ADT as neoadjuvant therapy for high-risk localized prostate cancer with IDC-P. The primary endpoint is the pathologic complete response (pCR).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically diagnosis of prostate cancer with positive IDC-P status
* High-risk localized prostate cancer, defined by either: Tumor stage ≥T3a by digital rectal examination, or Primary tumor Gleason score ≥ 8, or PSA > 20 ng/mL
* No evidence of metastases
* The ECOG score of the patient is ≤2
* Expected survival over 5 years
* Patients must participate voluntarily and sign an informed consent form (ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol
* Agree to collect the tumor tissue and blood samples needed for the research and apply them to related study
* Adequate hematologic, renal and hepatic function:

  * Absolute neutrophil count [ANC] ≥1.5 x 10^9/L
  * Platelet count [PLT] ≥100 x 10^9/L
  * Hemoglobin [HGB] ≥9 g/dL
  * Serum Total bilirubin [TBIL] ≤1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 2.5 x ULN
  * Serum albumin [ALB] ≥2.8 g/dL
  * Serum Creatinine ≤ 1.5 x ULN
  * Creatinine Clearance ≥ 40 mL/min

Exclusion Criteria:

* Prior androgen deprivation therapy (medical or surgical), radiation therapy or chemotherapy for prostate cancer
* Evidence of metastatic disease (M1) on imaging studies
* Pathological finding consistent with small cell, ductal or neuroendocrine carcinoma of the prostate
* Major surgery or severe trauma within 30 days before enrollment
* Patients with severe or uncontrolled concurrent，including but not limited to：

  * Severe or uncontrolled concurrent infections
  * Human immunodeficiency virus [HIV] infection positive
  * Suffer from acute or chronic active hepatitis B (HBsAg positive and HBV DNA>1x10^3/mL) Or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA>15 IU/mL)
  * Active tuberculosis, etc
* Abnormal cardiac function as manifested by NYHA (New York Heart Association) class III or IV heart failure，or clinically significant ventricular arrhythmias
* Uncontrolled hypertension（Systolic blood pressure≥160mmHg or Diastolic blood pressure≥100mmHg）
* Severe or unstable angina, myocardial infarction，arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks) Occurred within 6 months before enrollment
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Any condition that in the opinion of the investigator, would preclude participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patient can enter this study
Enrollment: 50 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate（pCR） | 6 months
  The proportion of subjects with no morphologically recognizable cancer cell in tumor specimens after radical prostatectomy.

SECONDARY OUTCOMES:
Rate of Subjects With Minimal Residual Disease | 6 months
  The proportion of subjects that have residual tumors with maximum diameter of 5 mm or less after radical prostatectomy.
Rate of positive surgical margin (PSM) | 6 months
  The rate of positive surgical margins in the prostatectomy specimen after neoadjuvant therapy.
Rate of Nodal Metastases After 6 Months of Treatment | 6 months
  The rate of the presence of tumor cells within surgically excised lymph nodes will be assessed after 6 months of neoadjuvant treatment.
Rate of Pathologic T3 Disease After 6 Months of Treatment | 6 months
  The rate of the presence of T3 disease (e.g. extraprostatic tumor not invading adjacent structures) will be determine from the prostatectomy specimen after 6 months of neoadjuvant treatment.
Biochemical Progression-free Survival (bPFS) | 2 years
  Biochemical progression will be defined per the American Urological Association guidelines (i.e. confirmed prostate-specific antigen post-radical prostatectomy >= 0.2 ng/mL) or death. Will be estimated using Kaplan-Meier methods and 95% CI will be estimated using Greenwood's formula.
PSA decline rate | 6 months
  The rate of PSA decline to baseline PSA after 6 months of neoadjuvant therapy.
Incidence and severity of adverse events | 6 months
  Safety as assessed by the incidence and severity of adverse events and serious adverse events graded according to the National Cancer Institute - Common Terminology Criteria for adverse events (CTCAE) version 4.0.
Quality of life (QOL) as assessed by FACT-P | Up to 24 months after surgery
  The QOL will be measured using the functional assessment of cancer therapy-prostate（FACT-P）. The questionnaires will be administered at baseline, prior to RP and every 3 months for 2 years post RP.
Quality of life as assessed by EQ-5D | Up to 24 months after surgery
  The QOL will be measured using the EuroQol five dimensions questionnaire（EQ-5D）. The questionnaires will be administered at baseline, prior to RP and every 3 months for 2 years post RP.
Radiographic progression-free survival (rPFS) | 2 years
  Time from surgery to radiographic progression or death
Overall survival | 5 years
  Time from surgery to death due to any cause

OTHER OUTCOMES:
Rate of Magnetic Resonance Imaging Downstaging after Neoadjuvant Therapy | 6 months
  The rate of MRI imaging downstaging after neoadjuvant therapy
Exploratory analysis to correlate tissue expression of PSA, CYP17, Ki67, and AR with pathologic response | 6 months
  To correlate the expression of PSA, CYP17, Ki67, and AR by immunohistochemistry with pCR/npCR in the prostatectomy specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zeng, Professor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Humphrey PA, Moch H, Cubilla AL, Ulbright TM, Reuter VE. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part B: Prostate and Bladder Tumours. Eur Urol. 2016 Jul;70(1):106-119. doi: 10.1016/j.eururo.2016.02.028. Epub 2016 Mar 17. PMID 26996659
- [Background] Efstathiou E, Abrahams NA, Tibbs RF, Wang X, Pettaway CA, Pisters LL, Mathew PF, Do KA, Logothetis CJ, Troncoso P. Morphologic characterization of preoperatively treated prostate cancer: toward a post-therapy histologic classification. Eur Urol. 2010 Jun;57(6):1030-8. doi: 10.1016/j.eururo.2009.10.020. Epub 2009 Oct 17. PMID 19853370
- [Background] Van der Kwast T, Al Daoud N, Collette L, Sykes J, Thoms J, Milosevic M, Bristow RG, Van Tienhoven G, Warde P, Mirimanoff RO, Bolla M. Biopsy diagnosis of intraductal carcinoma is prognostic in intermediate and high risk prostate cancer patients treated by radiotherapy. Eur J Cancer. 2012 Jun;48(9):1318-25. doi: 10.1016/j.ejca.2012.02.003. Epub 2012 Mar 8. PMID 22405699
- [Background] Kumar S, Shelley M, Harrison C, Coles B, Wilt TJ, Mason MD. Neo-adjuvant and adjuvant hormone therapy for localised and locally advanced prostate cancer. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD006019. doi: 10.1002/14651858.CD006019.pub2. PMID 17054269
- [Background] Zhao T, Liao B, Yao J, Liu J, Huang R, Shen P, Peng Z, Gui H, Chen X, Zhang P, Zhu Y, Li X, Wei Q, Zhou Q, Zeng H, Chen N. Is there any prognostic impact of intraductal carcinoma of prostate in initial diagnosed aggressively metastatic prostate cancer? Prostate. 2015 Feb 15;75(3):225-32. doi: 10.1002/pros.22906. Epub 2014 Oct 13. PMID 25307858
- [Background] Chen Z, Chen N, Shen P, Gong J, Li X, Zhao T, Liao B, Liu L, Liu Z, Zhang X, Liu J, Peng Z, Chen X, Xu M, Gui H, Zhang P, Wei Q, Zhou Q, Zeng H. The presence and clinical implication of intraductal carcinoma of prostate in metastatic castration resistant prostate cancer. Prostate. 2015 Sep;75(12):1247-54. doi: 10.1002/pros.23005. Epub 2015 Apr 27. PMID 25917338
- [Background] Zhao J, Shen P, Sun G, Chen N, Liu J, Tang X, Huang R, Cai D, Gong J, Zhang X, Chen Z, Li X, Wei Q, Zhang P, Liu Z, Liu J, Zeng H. The prognostic implication of intraductal carcinoma of the prostate in metastatic castration-resistant prostate cancer and its potential predictive value in those treated with docetaxel or abiraterone as first-line therapy. Oncotarget. 2017 Jul 24;8(33):55374-55383. doi: 10.18632/oncotarget.19520. eCollection 2017 Aug 15. PMID 28903426
- [Background] Porter LH, Lawrence MG, Ilic D, Clouston D, Bolton DM, Frydenberg M, Murphy DG, Pezaro C, Risbridger GP, Taylor RA. Systematic Review Links the Prevalence of Intraductal Carcinoma of the Prostate to Prostate Cancer Risk Categories. Eur Urol. 2017 Oct;72(4):492-495. doi: 10.1016/j.eururo.2017.03.013. Epub 2017 Mar 22. PMID 28342640
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] James ND, de Bono JS, Spears MR, Clarke NW, Mason MD, Dearnaley DP, Ritchie AWS, Amos CL, Gilson C, Jones RJ, Matheson D, Millman R, Attard G, Chowdhury S, Cross WR, Gillessen S, Parker CC, Russell JM, Berthold DR, Brawley C, Adab F, Aung S, Birtle AJ, Bowen J, Brock S, Chakraborti P, Ferguson C, Gale J, Gray E, Hingorani M, Hoskin PJ, Lester JF, Malik ZI, McKinna F, McPhail N, Money-Kyrle J, O'Sullivan J, Parikh O, Protheroe A, Robinson A, Srihari NN, Thomas C, Wagstaff J, Wylie J, Zarkar A, Parmar MKB, Sydes MR; STAMPEDE Investigators. Abiraterone for Prostate Cancer Not Previously Treated with Hormone Therapy. N Engl J Med. 2017 Jul 27;377(4):338-351. doi: 10.1056/NEJMoa1702900. Epub 2017 Jun 3. PMID 28578639